CLINICAL TRIAL: NCT06280612
Title: The Effect of Live Cat and Simulation Cat Therapies on Oncology Patients' Post-Chemotherapy Symptoms and Happiness Levels: A Randomized Controlled Study
Brief Title: The Effect of Live Cat and Simulation Cat Therapies on Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Hatice Demirağ, Ph.D, Asst. Prof., Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RCS10042023
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Therapy-Associated Cancer; Cancer Patient; Happiness; Symptoms
Keywords: pet therapy; cancer patient; happiness; symptoms
MeSH Terms: conditions — Neoplasms, Second Primary | interventions — Animal Assisted Therapy

STUDY DESIGN:
Intervention Model Description: The sample number of the research was calculated in the G*Power 3.1.9.6 program. While α=0.05 was the error amount, 0.628 was the effect size, and 0.90 (90%) was the targeted test power, it was calculated as 36 patients for three groups (living cat group, robotic cat group, control group). Since there was no previous study on the subject, a study examining happiness levels in a different sample group was used as a reference. Considering situations such as wanting to leave the study or death during the research, each group was increased by 25%, and a total of 45 patients, 15 patients for each group, were included in the study.
Who Masked: Participant
Masking Description: Since the possibility of patients being affected by each other was minimal, the study was continued with only one of the live cat groups, the simulation cat group, and the control group. For example, only the live cat group and those who received chemotherapy treatment were studied before Monday afternoon.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Live Cat Group (Experimental): Before starting the study, the "Structured Patient Information Form," "Edmonton Symptom Diagnosis Scale," and "Oxford Happiness Scale Short Form" were applied to the patients. Then, the researcher gave the patients face-to-face, individual information about hand hygiene after contact with a live cat for approximately 15 minutes in the waiting room and offered them a "Live Cat Information Brochure." Patients were then asked to spend 20 minutes with a pet at home twice a week for 12 weeks. "Edmonton Symptom Diagnosis Scale" and "Oxford Happiness Scale Short Form" were applied to this group of patients three times: before, at the 6th week, and at the end of the 12th week of the study.
  Interventions: Other: Pet therapy
- Robotic Cat Group (Experimental): Before starting the study, the "Structured Patient Information Form," "Edmonton Symptom Diagnosis Scale," and "Oxford Happiness Scale Short Form" were applied to the patients. Then, the researcher gave the patients face-to-face information about the robotic cat "Silver" and its use for approximately 15 minutes in the waiting room and offered them a "Robotic Cat Information Brochure." In each pet therapy application, patients' hand hygiene and cleaning of the Robotic Cat was provided, the robot cat was given to the patients.
  Interventions: Other: Pet therapy
- Control Group (No Intervention): Before starting the study, the "Structured Patient Information Form", "Edmonton Symptom Diagnosis Scale", and "Oxford Happiness Scale Short Form" were applied to the patients. Treatment was given to this group of patients only after informing them about the study, and the patients were followed for only three months. "Edmonton Symptom Diagnosis Scale" and "Oxford Happiness Scale Short FormS" were applied to the patients three times: before, at the 6th week, and the end of the 12th week of the research.

INTERVENTIONS:
Other: Pet therapy — The patients were allowed to spend time with an animal (cat/robotic cat) for 20 minutes twice a week for 12 weeks.
  Arms: Live Cat Group; Robotic Cat Group

SUMMARY:
It is known that animals are good for humans physiologically and psychologically. Therefore, in this study, the effects of live cat and robotic cat therapies on the symptoms and happiness levels of oncology patients after chemotherapy were examined.

DETAILED DESCRIPTION:
Cancer is a disease that requires a long-term struggle with the psychosocial and economic burden it creates on the individual, family and society, bringing with it many health problems. Although chemotherapy treatment is the main treatment method for patients, it can cause some changes in the individual's appearance while treating cancer and many symptoms such as nausea, vomiting, diarrhea, alopecia, and constipation after treatment. At the same time, patients may feel tired, sleepy and depressed after treatment. However, cancer patients and their families experiencing some unknown diagnosis and treatment processes related to cancer also cause them to be unhappy as a result of experiencing some physical, social, emotional and spiritual problems during the treatment.

It is reported in the literature that pet therapy or animal-assisted treatments reduce disease-related symptoms and make patients happy. Pet therapy is an auxiliary non-pharmacological form of treatment that heals physiological and psychological diseases through interactions between animals and humans that meet certain criteria, and stimulates and activates the body mechanisms required for the development of the individual's health behaviors. In the literature, pet therapy studies with oncology patients are quite limited. Therefore, this study was conducted to examine the effects of live cat and robotic cat therapies on the symptoms and happiness levels experienced by oncology patients after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for admission to the study are 18≤ of age,
* Agreeing to participate in the research,
* Being conscious of receiving outpatient chemotherapy treatment for 3≤ months, and being able to communicate.
* The criteria included no impairment in mental and cognitive functions of patients/relatives in the live group,
* Patients in the live cat group not having any animal allergies, and the cat group having a cat.

Exclusion Criteria:

* Not agreeing to participate in the research,
* Being under 18 years of age,
* Having known psychological disorders, having a visual, hearing, or speech disability, and having an animal allergy.
* Also excluded are having a surgical wound (suture, drainage, etc.), neutropenia or severe infection (by resistant bacteria), fever, diarrhea, respiratory symptoms or vomiting during the week before the start of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Edmonton Symptom Diagnostic Scale | 12 Weeks
  The scale includes "pain, fatigue, nausea, sadness, anxiety, insomnia, loss of appetite, the feeling of well-being, shortness of breath and other problems (changes in the skin and nails, sores in the mouth, numbness in the hands)." Sadırlı and Ünsar added other problems to the scale. Therefore, the current version with 11 items was used in this study. The severity of each symptom ranges from "no symptoms" to "very severe," with increasing numerical intensity between 0 and 10.
  "Edmonton Symptom Diagnostic Scale" were administered to the patients three times in total before the study (pretest), at the sixth week/middle (intermediate measurement), and the end of the 12th week/end of the survey (posttest).
Oxford Happiness Scale Short Form | 12 Weeks
  In the Turkish adaptation, the scale has seven items and a 5-point Likert type. The scores obtained from the items on the scale vary from "1 point: I Completely Disagree" to "5 points: I Completely Agree", with the lowest being seven and the highest being 35 points.
  "Oxford Happiness Scale Short Form" were administered to the patients three times in total before the study (pretest), at the sixth week/middle (intermediate measurement), and the end of the 12th week/end of the survey (posttest).

CONTACTS AND LOCATIONS:
Locations (1):
- Gümüşhane University, Gümüşhane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I'll decide later